CLINICAL TRIAL: NCT02303080
Title: Whey Protein Micelles and Thermogenesis In Overweight Subjects
Acronym: Thermowhey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 10.19.MET
Record Dates: First submitted 2014-11-10; First posted 2014-11-27 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2014-11

CONDITIONS: Overweight
Keywords: whey protein microgels; thermogenesis
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (WPM 0) (Placebo Comparator): 400 mL beverage with 85.0% maltodextrine, 15.0% fat and 0% of whey protein micelles Product given once after 1 hour of monitoring for baseline
  Interventions: Other: WPM 30; Other: WPM 50; Other: MC 50
- WPM 30 (Active Comparator): 400 mL beverage with 43.7% of maltodextrine, 15.2 % fat and 41.1% (30 g) of whey protein micelles Product given once after 1 hour of monitoring for baseline
  Interventions: Other: Control (WPM 0); Other: WPM 50; Other: MC 50
- WPM 50 (Active Comparator): 400 mL beverage with 16.3% of maltodextrine, 15.2 % fat and 68.5% (50 g) of whey protein micelles Product given once after 1 hour of monitoring for baseline
  Interventions: Other: Control (WPM 0); Other: WPM 30; Other: MC 50
- MC 50 (Active Comparator): 400 mL beverage with 16.7% of maltodextrine, 15.0 % fat and 68.2% (50 g) of whey protein micelles 50 g of micellar casein Product given once after 1 hour of monitoring for baseline
  Interventions: Other: Control (WPM 0); Other: WPM 30; Other: WPM 50

INTERVENTIONS:
Other: Control (WPM 0) — 85.0 % maltodextrin,15.0% fat, 0% WPM
  Arms: MC 50; WPM 30; WPM 50
Other: WPM 30 — 43.7% maltodextrin, 15.2% fat, 41.1% (30 g) WPM
  Arms: Control (WPM 0); MC 50; WPM 50
Other: WPM 50 — 16.3% maltodextrin, 15.2% fat, 68.5% (50 g) WPM
  Arms: Control (WPM 0); MC 50; WPM 30
Other: MC 50 — 16.7% maltodextrin, 15.0% fat, 68.2% (50 g) MC
  Arms: Control (WPM 0); WPM 30; WPM 50

SUMMARY:
The main objective of the trial is to measure the thermogenic effect of two different doses of whey protein microgels.

It will be a randomized crossover double-blind design conducted in 20 subjects.

DETAILED DESCRIPTION:
Primary objective and outcome:

The primary objective of the trial is to measure the thermogenic effect of two different doses of whey protein microgels (WPM).

Secondary objectives and outcomes:

Explore the mechanism of action of WPM on thermogenesis including:

Protein turnover in response to the dose and the source of protein (WPM versus casein) Insulinemic and glycemic response to the dose and source of protein (WPM versus casein)

Design: The proposed study is a randomized double-blind, placebo-controlled, single center, crossover design.

At the start of the study, subjects will be randomly assigned to 4 different groups in a crossover design, where they will be asked to consume a beverage containing Product 1: 0g of protein (maltodextrin control) Product 2: 30g of WPM Product 3: 50g of WPM Product 4: 50g of micellar casein (MC) Number of subjects: The number of subjects will be 15. Sufficient subjects should be recruited to provide a 30% drop-out rate. Therefore 20 subjects will be needed including drop-outs.

ELIGIBILITY:
Inclusion Criteria:

Overweight (BMI range between 25.0 and 29.9 kg per m2 Healthy Having obtained his/her subjects over 20 year informed consent.

Exclusion Criteria:

Chronic or acute diseases affecting protein metabolism (diabetes, renal insufficiency, CVD, liver disease), dyslipidemia History of varicose or venous stases Recent major surgery (3 months) History of major gastro-intestinal surgery (gastric bypass, intestinal resection etc…) Malabsorption disorders History of cancer within the past year Significant weight loss during the last 3 months Food allergies, especially cow milk protein. Pregnancy or lactation Special diets especially vegetarian, high protein (≥ 1.6 g/kg) or weight loss program Abnormal Food Frequency Questionnaire Aversion to vanilla or chocolate aromas Smoking Moderate to intense physical activity > 2 hours/week Hematocrit <40 for males and < 36 for females Blood donation within 3 months of study start and 3 months after study end Regular consumption of medication and supplements i.e. any treatment affecting thermogenesis or nutrient metabolism in general such as corticosteroids, insulin, androgens, antibiotics and nutritional supplements (multivitamins, protein shakes).

Have a high alcohol consumption (more than 1 drink/day) Consumption of illicit drugs Subject who cannot be expected to comply with the study procedures, including consuming the test products.

Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
thermic effect of food | 7 hours from baseline measurements
  gas exchanges through indirect calorimetry

SECONDARY OUTCOMES:
Whole body protein turnover | 7 hours from baseline
  protein synthesis and breakdown

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD, PhD, Principal Investigator — Société des Produits Nestlé (SPN)

REFERENCES:
- [Derived] Kassis A, Godin JP, Moille SE, Nielsen-Moennoz C, Groulx K, Oguey-Araymon S, Praplan F, Beaumont M, Sauser J, Monnard I, Kapp AF, Ammon-Zufferey C, Frei N, Guignard L, Delodder F, Mace K. Effects of protein quantity and type on diet induced thermogenesis in overweight adults: A randomized controlled trial. Clin Nutr. 2019 Aug;38(4):1570-1580. doi: 10.1016/j.clnu.2018.08.004. Epub 2018 Aug 10. PMID 30269898